CLINICAL TRIAL: NCT05491772
Title: Clasificación y Factores de Riesgo de la Mortalidad Perinatatal
Brief Title: Multicentric Retrospective Study of Perinatal Mortality
Acronym: PM-PHD-NTM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Hospital Sant Joan de Deu (Other); Hospital Clínic Sede Maternitat (Other)
Responsible Party: Principal Investigator, Nuria Torre-Monmany, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: Perinatal mortality - pHD NTM
Record Dates: First submitted 2022-07-24; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Perinatal Morbidity; Morbidity;Perinatal; Stillbirth; ICD
Keywords: perinatal mortality; ICD; Perinatal death; stillbirth; neonatal mortality; cause of death; risk factors
MeSH Terms: conditions — Stillbirth; Perinatal Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Perinatal mortality ranges mortality from 22 gestational weeks up to the first 7 days of life and extended mortality goes up to 28 days of life. The perinatal mortality rate is the most sensitive index of the health status of women and their offspring and of the quality of maternal and child health services. Per our knowledge, there is no study that evaluates perinatal mortality in Catalonia, although household data are available from each hospital. Moreover, the official records usually do not match with the household surveys due to lack of clarity on the definitions. Aim: the aim of the study is to compare the WHO perinatal mortality classification following the ICD-PM in comparison with the used classification. Methodology: Multicentric retrospective study. Data from Sant Joan de Déu, Maternitat Clinic and Parc Taulí hospitals.

ELIGIBILITY:
Inclusion Criteria:

* stillbirths more than 22 weeks of gestation
* neonatal deaths up to 28 days of life

Exclusion Criteria:

- avortions more than 22 weeks of gestation

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Perinatal
Sampling Method: Non-Probability Sample
Enrollment: 468 (Estimated)
Dates: Start 2022-08-05 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
International Classification of Disease (10th Revision)- Perinatal Mortalitymaternal condition group | through study completion, an average of 1 year
  The ICD-PM provides a standardised system for classifying perinatal mortality (including stillbirths) based on time of death (antepartum or intrapartum) into fetal and maternal causes thereby enabling comparisons within and between diverse settings and contexts
International Classification of Disease (10th Revision)- Perinatal Mortality cause of death | through study completion, an average of 1 year
  The ICD-PM provides a standardised system for classifying perinatal mortality (including stillbirths) based on time of death (antepartum or intrapartum) into fetal and maternal causes thereby enabling comparisons within and between diverse settings and contexts

SECONDARY OUTCOMES:
Obstetric history | through study completion, an average of 1 year
  number of pregnancies, number of total live births, number of deceased babies, number of stillbirths, number of neonatal deaths, number of abortions
Mother's age | through study completion, an average of 1 year
  age
Type of pregnancy | through study completion, an average of 1 year
  singleton, twins
Antenatal care number of visits | through study completion, an average of 1 year
  number
Malaria profilaxis | through study completion, an average of 1 year
  yes, no
HIV status | through study completion, an average of 1 year
  positive, negative
Syphilis test | through study completion, an average of 1 year
  positive, negative
Mother's LMP | through study completion, an average of 1 year
  date of the last menstrual period
Date of birth | through study completion, an average of 1 year
  date
Gestational age | through study completion, an average of 1 year
  weeks
Place of delivery | through study completion, an average of 1 year
  facility, home, road, others
Onset of labour | through study completion, an average of 1 year
  spontaneous, induced, cesarean before onset
Fetal heart sounds on admission | through study completion, an average of 1 year
  yes, no
Partograph used | through study completion, an average of 1 year
  yes, no
Mode of delivery | through study completion, an average of 1 year
  vaginal, vaginal assisted, cesarean
Time between decision for action and birth | through study completion, an average of 1 year
  not applicable, < 30 min, 30 - 60 min, > 60 min
Apgar Score | through study completion, an average of 1 year
  Apgar Score (min 0, max 10). Higher scores means better outcome
Resuscitation | through study completion, an average of 1 year
  not necessary, suction, stimulation, ventilation, cardiac compressions, not done
Sex of baby | through study completion, an average of 1 year
  male, female, unknown
Birth weight | through study completion, an average of 1 year
  grams
Date of death | through study completion, an average of 1 year
  Date
Type of death | through study completion, an average of 1 year
  neonatal, intrapartum or antepartum or unknown timing stillbirth

CONTACTS AND LOCATIONS:
Locations (1):
- CorporacionPT, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torre Monmany N, Astete JA, Ramaiah D, Suchitra J, Krauel X, Fillol M, Balasubbaiah Y, Alarcon A, Bassat Q. Extended Perinatal Mortality Audit in a Rural Hospital in India. Am J Perinatol. 2023 Mar;40(4):375-386. doi: 10.1055/s-0041-1727220. Epub 2021 Apr 26. PMID 33902133